CLINICAL TRIAL: NCT02530710
Title: A Phase 1, Randomized, Placebo-Controlled, Double-Blind, Dose-Escalation Study to Evaluate Safety, Tolerability and Pharmacokinetics of Single Doses of Q203 in Normal, Healthy, Male and Female Volunteers
Brief Title: A Dose-Escalation Study to Evaluate Safety, Tolerability and Pharmacokinetics of Single Doses of Q203 in Normal, Healthy, Male and Female Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Qurient Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Q203-TB-PI-US001
Record Dates: First submitted 2015-08-18; First posted 2015-08-21 (Estimated); Last update posted 2016-12-06 (Estimated); Status verified 2016-08

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — telacebec

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Q203 (Experimental): Q203 drug products (10mg and 100mg tablets)
  Interventions: Drug: Q203
- Placebo (Placebo Comparator): Placebo tablets (same excipients used in Q203 drug products)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Q203
  Arms: Q203
Drug: Placebo
  Arms: Placebo

SUMMARY:
Randomized, double-blind, placebo-controlled, dose-escalation study in healthy male and female volunteers. Subjects will be randomly assigned to 1 of 7 treatment cohorts (Cohorts 1 - 7) of 8 subjects each, to receive either Q203 or placebo (6 active treatment : 2 placebo) in a fasting state.

Dose escalation to the next cohort may be considered when at least 6 out of 8 subjects, in a cohort, completes all procedures and none of the subjects has a clinically significant adverse event (AE) that is being followed, or at the discretion of the PI if no drug-related serious adverse events (SAEs) have occurred.

A food effect cohort will be enrolled to test administration of Q203 in a fed state, at 100 mg dose level (this dose level may change based on PK analysis results). Subjects who received 100mg dose in a fasting state will return and receive the second dose, with food.

Subjects will be followed up for AEs, SAE or pregnancy for 30 days postdrug administration.

DETAILED DESCRIPTION:
Randomized, double-blind, placebo-controlled, dose-escalation study in healthy male and female volunteers. Subjects will be randomly assigned to 1 of 7 treatment cohorts (Cohorts 1 - 7) of 8 subjects each, to receive either Q203 or placebo in a fasting state. Every attempt will be made to include at least 2 females in each cohort, at least one of whom will be assigned to receive Q203.

Dose escalation to the next cohort may be considered when at least 6 out of 8 subjects, in a cohort, completes all procedures and none of the subjects has a clinically significant adverse event (AE) that is being followed, or at the discretion of the PI if no drug-related SAEs have occurred. A food effect cohort will be enrolled to test administration of Q203 in a fed state, at 100 mg dose level (this dose level may change based on PK analysis results). Subjects who received 100mg dose in a fasting state will return and receive the second dose, with food. In this cohort, all eight subjects will proceed to receive either Q203 or placebo in a six to two ratio (six active treatment : 2 placebo). Every attempt will be made to include at least 2 females in this cohort, at least one of whom will be assigned to receive Q203.

Subjects will be followed up for AEs, SAE or pregnancy for 30 days postdrug administration.

ELIGIBILITY:
Inclusion Criteria:

1. Able to understand and sign an informed consent form.
2. Healthy adult males and females of non-childbearing potential, ages 18 to 55 years, inclusive at the time of screening.
3. Body mass index of 18 to 32 kg/m2, inclusive, and weighing at least 50 kg.
4. Female subjects must be of non-childbearing potential (postmenopause or surgical sterilization). Postmenopausal status will be confirmed by a follicle-stimulating hormone (FSH) test at screening.
5. Male subjects must agree to use a condom with spermicide when engaging in sexual intercourse during the study period and for 30 days after study drug dosing, if they have not had a vasectomy at least 6 months before study start.
6. Male subjects must not donate sperm during the study and for 30 days after study drug dosing.
7. Able to understand and comply with all of the study requirements.
8. Able to swallow 8 tablets in succession.
9. Willing to fast a minimum of 8 hours before check-in.
10. Agree not to donate blood, plasma, platelets or any other blood components for 1 month after receiving study drug.
11. Willing to abstain from alcohol use from 48 hours before check-in through the end of the study.
12. Willing to forgo sunbathing and prolonged exposure to sunlight during the study period.
13. Willing to forgo strenuous exercise during the study period.

Exclusion Criteria:

1. Any known chronic systemic viral infection (including a positive serological test for HIV, HBsAg or HCAb that indicates infection).
2. History of or current active tuberculosis (TB).
3. Any systemic infection or other systemic illness, including persistent cough, respiratory, or flu-like symptoms, in the previous 30 days before screening.
4. History of histoplasmosis, coccidioidomycosis, or similar opportunistic fungal infection.
5. Vaccination in the previous 30 days before screening.
6. History of, or clinically significant evidence of, bradycardia, syncope, or ECG abnormality or any other cardiovascular abnormality.
7. Resting heart rate (HR) during screening or baseline ECG fewer than 50 beats per minute (bpm).
8. History of seizures.
9. History of drug (including amphetamines, barbiturates, benzodiazepines, cocaine, opiates, phencyclidines, and cannabinoids) or alcohol abuse or addiction within the past 2 years or, if male, consumes more than 28 units of alcohol per week or, if female, consumes more than 21 units of alcohol per week (1 unit of alcohol equals 250 mL of beer, 100 mL of wine, or 25 mL of spirits).
10. Any history of abnormal pulmonary function (e.g., asthma or related respiratory illnesses).
11. Current or recent (within the past 3 months) use of tobacco or other nicotine-containing product or positive results for nicotine testing at screening or check-in.
12. Use of any prescription or over-the-counter (OTC) drug or herbal product within 14 days before dosing.
13. Use of any known drug metabolism enzyme-altering drug (inducers or inhibitors) or supplement (e.g., St. John's wort) within 14 days before dosing or consumption of foods or beverages containing alcohol or grapefruit within 48 hours before dosing.
14. Use of any QT-prolonging agents, including, but not limited to, azithromycin, bepridil chloroquine, chlorpromazine, cisapride, clarithromycin, disopyramide dofetilide, domperidone, droperidol, erythromycin, Halofantrine, haloperidol, ibutilide, levomethadyl, lumefantrine, mefloquine, mesoridazine, methadone, moxifloxacin, pentamidine, pimozide, procainamide, quinidine, quinine, roxithromycin, sotalol, sparfloxacin, terfenadine, or thioridazine, from within 28 days before dosing through end of study.
15. Any prior exposure to Q203 or participation in another investigational drug study within the previous 30 days before screening.
16. Any donation of blood, plasma, or platelets or significant loss of blood within 56 days before dosing.
17. Laboratory results outside the normal range, if considered clinically significant by the PI or his designee.
18. Hemoglobin concentration < LLN.
19. Any condition that might interfere with the absorption of the study medications.
20. History of hypersensitivity or idiosyncratic reaction to any of the products administered during the study.
21. History of unexplained syncope or fainting from the collection of blood, i.e., autonomic dysfunction.
22. History of hypotension, including orthostatic hypotension.
23. Inability to understand verbal and/or written English.
24. Subjects with glucose-6-phosphate-dehydrogenase (G6PD) deficiency.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 56 (Actual)
Dates: Start 2015-08; Primary Completion 2016-01 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Safety assessed through adverse events, vital signs, ECG, laboratory results, and telemetry monitoring | 7 days post dose

SECONDARY OUTCOMES:
Pharmacokinetic analysis: Area under the plasma concentration | predose and 1, 2, 4, 5, 6, 8, 12, 24, 48, 72, 96, 120, 144, 216 and 312 hours postdose
Pharmacokinetic analysis: Maximum observed plasma drug concentration | predose and 1, 2, 4, 5, 6, 8, 12, 24, 48, 72, 96, 120, 144, 216 and 312 hours postdose
Pharmacokinetic analysis: Time of maximum observed concentration | predose and 1, 2, 4, 5, 6, 8, 12, 24, 48, 72, 96, 120, 144, 216 and 312 hours postdose

CONTACTS AND LOCATIONS:
Locations (1):
- Baltimore, Maryland, United States